CLINICAL TRIAL: NCT02833766
Title: Anti-EGFR-immunoliposomes Loaded With Doxorubicin in Patients With Advanced Triple Negative EGFR Positive Breast Cancer - A Multicenter Single Arm Phase II Trial
Brief Title: Anti-EGFR-immunoliposomes Loaded With Doxorubicin in Patients With Advanced Triple Negative EGFR Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the trial was prematurely terminated as per SAKK board decision from 14th of November 2020. The trial is to be terminated after primary endpoint is reached.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 24/14
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; advanced triple Negative, EGFR positive breast cancer; doxorubicin; triple negative breast cancer (TNBC)
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- anti-EGFR-IL-dox (Experimental): Metastatic, non resectable, EGFR positive TNBC patients treated in first-line
  Interventions: Drug: anti-EGFR-IL-dox

INTERVENTIONS:
Drug: anti-EGFR-IL-dox — First-line treatment with anti-EGFR-IL-dox, given at a dose of 50 mg/m2 intravenous, on day 1 of each cycle, cycle length is 28 days
  Other Names: anti-EGFR-immunoliposomes loaded with doxorubicin

SUMMARY:
The main objective of the trial is to determine the efficacy of doxorubicin-loaded anti-EGFR immunoliposomes as first-line therapy in patients with advanced triple Negative, EGFR positive breast cancer. In this proof of concept trial, all patients will have an administration of the doxorubicin-loaded anti-EGFR immunoliposomes (anti-EGFR-IL-dox) every 28 days, until progression or unacceptable toxicity.

DETAILED DESCRIPTION:
Advanced triple negative breast cancer (TNBC) is a highly chemosensitive disease displaying a dismal short-term prognosis with more than three quarters of patients in progression 12 months after the initiation of conventional chemotherapy. Approximately 2/3 of TNBC are expressing EGFR and breast cancer, including TNBC, is a disease highly sensitive to anthracyclines. Furthermore, data from a phase I trial, in 26 patients with different solid tumors, show very little toxicity and signs of efficacy of anti-EGFR-IL-dox.

The EGFR assessment will be performed centrally and only patients with EGFR positive tumors will be included. The patients will be treated with the anti-EGFR-IL-dox until progression and followed-up according to standard practice for patient with TNBC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before prescreening and registration and prior to any trial specific procedures, including participation in mandatory translational research
* Histologically proven diagnosis of TNBC in metastatic or locally advanced non operable stage
* EGFR expression in primary tumor or metastases of at least (1+) in immunohistochemistry, assessed by central pathologist
* Measurable or evaluable disease according to RECIST 1.1
* No prior systemic treatment for metastatic or inoperable disease
* Adequate bone marrow function: neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L
* Adequate hepatic function: total bilirubin ≤ 1.5 x ULN; AST, ALT and AP ≤ 2.5 x ULN (AST, ALT and AP ≤ 5 x ULN if hepatic metastases are the only reason for enzyme elevation)
* Adequate renal function: serum creatinine ≤ 1.5 x ULN and calculated creatinine clearance > 30 mL/min, according to the formula of Cockcroft-Gault.
* Adequate cardiac function: Left Ventricular Ejection Fraction (LVEF) ≥ 40% as determined by either echocardiography (ECHO) or radionuclide angiocardiography (MUGA)

Exclusion Criteria:

* Evidence of CNS or leptomeningeal metastases (even if previously treated); CNS imaging not required in asymptomatic patients
* History of hematologic or primary solid tumor malignancy, unless in remission for at least 5 years from registration. Inclusion of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer is permitted independent of time since diagnosis
* Previous therapy with more than 240 mg/m2 of doxorubicin or more than 450 mg/m2 of epirubicin
* Previous radiotherapy for the metastatic disease (palliative radiotherapy of only non-target lesions is allowed)
* Adjuvant treatment must have been stopped at least 6 months before registration
* Any serious underlying medical condition (at the judgement of the investigator) which could impair the ability of the patient to participate in the trial (e.g. active autoimmune disease, uncontrolled diabetes, etc.)
* Breastfeeding
* Participation in any investigational drug trial within 4 weeks preceding treatment start
* Any concomitant drugs contraindicated when administering Erbitux™ or Caelyx™ according to the Swissmedic-approved product information
* Known hypersensitivity to trial drug(s) or to any component of the trial drug(s)
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | at 12 months after registration
  PFS is defined as the time from registration until progression according to RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | at 12 months after registration
  ORR is defined as proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 during trial treatment.
Duration of response (DOR) | at 12 months after registration
  DOR is defined as time from the date when a patient first meets the criteria for CR or PR according to RECIST v1.1, until documented progression, relapse or death due to disease progression, whichever occurs first.
Time to Progression (TTP) | at 12 months after registration
  Time to Progression (TTP), defined as the time from registration until progression TTP assessed according to RECIST v1.1 or death due to disease progression, whichever occurs first.
PFS | at 12 months after registration
  PFS is defined as the time from registration until progression according to RECIST v1.1 or death from any cause, whichever occurs first.
Overall survival (OS) | at 12 months after registration
  OS is defined as time from registration until death from any cause.
Adverse events (AEs) | at 12 months after registration
  AE are assessed according to NCI CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Winterhalder, MD, Study Chair — Luzerner Kantonsspital
Locations (15):
- Switzerland (15):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Inselspital, Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Hôpital de Sion, Sion
  - Spital STS AG, Thun
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum - Klinik im Park, Zurich
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mamot C, Wicki A, Hasler-Strub U, Riniker S, Li Q, Holer L, Bartschi D, Zaman K, von Moos R, Dedes KJ, Boos LA, Novak U, Bodmer A, Ritschard R, Obermann EC, Tzankov A, Ackermann C, Membrez-Antonioli V, Zurrer-Hardi U, Caspar CB, Deuster S, Senn M, Winterhalder R, Rochlitz C. A multicenter phase II trial of anti-EGFR-immunoliposomes loaded with doxorubicin in patients with advanced triple negative breast cancer. Sci Rep. 2023 Mar 6;13(1):3705. doi: 10.1038/s41598-023-30950-z. PMID 36879012